CLINICAL TRIAL: NCT06602128
Title: The Effect of Breathing Exercise on Anxiety, Pain and Vital Signs in Patients Undergoing Coronary Angiography: A Randomised Controlled Study
Brief Title: The Effect of Breathing Exercise on Anxiety, Pain and Life Findings in Patients Undergoing Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaraş İstiklal University (Other)
Responsible Party: Principal Investigator, Yasemin Sazak, Assistant Professor, Kahramanmaraş İstiklal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstiklalU-YSazak-001
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Breathing Exercises; Coronary Angiography
Keywords: Vital Signs; Pain; Stress
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The post-test measurements will be collected by a nurse working in the angiography ward who is not connected with the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercise Application Group (Experimental): Patients in the breathing exercise practice group will have breathing exercise practice for 15-20 minutes half an hour before the angiography procedure. The breathing exercise application will be applied to the patients face to face by the researcher.
  Interventions: Behavioral: Experimental: Breathing Exercise Application Group
- Control group (No Intervention): There will be no intervention for individuals in this group.

INTERVENTIONS:
Behavioral: Experimental: Breathing Exercise Application Group — The Effect of Breathing Exercise on Anxiety, Pain and Life Findings in Patients Undergoing Coronary Angiography
  Arms: Breathing Exercise Application Group

SUMMARY:
This randomised controlled trial will be conducted to evaluate the effect of breathing exercise on anxiety, pain and vital signs in patients undergoing coronary angiography before angiography.

Hypotheses of the study; H11: The anxiety level of the patients who underwent breathing exercise is lower than the patients in the control group.

H12: The pain level of the patients who underwent breathing exercise is lower than the control group H13: The vital signs of the patients who underwent breathing exercises are within normal limits compared to the control group.

In the study, there will be an intervention group in which breathing exercise will be applied and a control group in which no intervention will be applied.

Data will be collected with the pre-test data collection form half an hour before the angiography procedure in patients in the intervention and control groups. Patients in the intervention group will be given breathing exercises, while patients in the control group will not be subjected to any intervention. After the angioplasty procedure, data will be collected from the intervention and control groups with post-test data collection forms.

DETAILED DESCRIPTION:
In determining the groups; simple randomisation method will be used in order to form the sample in a way to ensure equal number and random distribution of the two groups. Randomisation will be done by using the website (https://www.randomizer.org). In line with the randomisation list; patients who meet the inclusion criteria will be included in the intervention and control groups. Inclusion in the intervention and control groups will be made by the researchers in line with the randomisation list. In order for the responsible researcher to apply breathing exercises; he/she has a breathing techniques coaching certificate. In the research; triple breathing technique (full yogic breathing) and square breathing technique will be used. Patients will be informed about the research and their written and verbal consent will be obtained. Data will be collected with the pre-test data collection form half an hour before the angiography procedure in patients in the intervention and control groups. Patients in the intervention group will be given breathing exercises, while patients in the control group will not be subjected to any intervention. The breathing exercise will be performed as a single session and will last approximately 15-20 minutes. After the angioplasty procedure, data will be collected from the intervention and control groups with post-test data collection forms.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary angiography for the first time
* Over 18 years of age
* No respiratory distress
* No problems with communication
* Volunteering to be included in the study.

Exclusion Criteria:

* Taking any medication to suppress anxiety symptoms
* Patients undergoing emergency coronary angiography and/or patients complaining of chest pain
* Patients on antihypertensive treatment before the procedure due to hypertension
* Patients who underwent emergency intervention during coronary angiography, surgical procedure and intensive care unit for follow-up were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Vital Signs Recording Form-Blood pressure values | 30 minutes before coronary angiography
  It is a form created by the researcher in which the blood pressure values of the patients are recorded.
Vital Signs Recording Form-Blood pressure values | Within 15 minutes after the angiography procedure is completed and the patient is taken to bed
  It is a form created by the researcher in which the blood pressure values of the patients are recorded.
Vital Signs Recording Form- Saturation | 30 minutes before coronary angiography
  It is a form created by the researcher in which the saturation values of the patients are recorded.
Vital Signs Recording Form- Saturation | Within 15 minutes after the angiography procedure is completed and the patient is taken to bed
  It is a form created by the researcher in which the saturation values of the patients are recorded.
Vital Signs Recording Form- Pulse values | 30 minutes before coronary angiography
  It is a form created by the researcher in which the pulse rates of the patients are recorded.
Vital Signs Recording Form- Pulse values | Within 15 minutes after the angiography procedure is completed and the patient is taken to bed
  It is a form created by the researcher in which the pulse rates of the patients are recorded.
Visual Analogy Scale (VAS) | 30 minutes before coronary angiography
  It is a 10 cm ruler that reflects the minimum and maximum state of pain by using it horizontally or vertically. '0' indicates painlessness and "10" indicates the most severe pain. The patient marks the intensity of pain felt on this ruler.
Visual Analogy Scale (VAS) | Within 15 minutes after the angiography procedure is completed and the patient is taken to bed
  It is a 10 cm ruler that reflects the minimum and maximum state of pain by using it horizontally or vertically. '0' indicates painlessness and "10" indicates the most severe pain. The patient marks the intensity of pain felt on this ruler.
State-Trait Anxiety Inventory (STAI-I) | 30 minutes before coronary angiography
  The scale developed by Spielberg et al. (1964) was adapted into Turkish by Öner and Le Compte (1974-1977). The reliability of the scale is determined between 0.83 and 0.92 and it requires the person to understand his/her situation at certain times and conditions and to mark one of the preferences '1 (Not at all), 2 (A little), 3 (Very), 4 (Completely)' according to its severity. The total score obtained from the scale varies between 20-80 and 20-39 indicates mild anxiety level, 40-59 indicates moderate anxiety level, 60-79 indicates high anxiety level and 80 points indicates panic anxiety level.
State-Trait Anxiety Inventory (STAI-I) | Within 15 minutes after the angiography procedure is completed and the patient is taken to bed
  The scale developed by Spielberg et al. (1964) was adapted into Turkish by Öner and Le Compte (1974-1977). The reliability of the scale is determined between 0.83 and 0.92 and it requires the person to understand his/her situation at certain times and conditions and to mark one of the preferences '1 (Not at all), 2 (A little), 3 (Very), 4 (Completely)' according to its severity. The total score obtained from the scale varies between 20-80 and 20-39 indicates mild anxiety level, 40-59 indicates moderate anxiety level, 60-79 indicates high anxiety level and 80 points indicates panic anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Sevinç Meşe, Study Chair — Kahramanmaraş İstiklal University
Locations (1):
- Kahramanmaraş Istiklal Universty, Kahramanmaraş, Turkey (Türkiye)